CLINICAL TRIAL: NCT06717815
Title: A Multi-center, Multi-dose Phase Ib/IIa Clinical Study Evaluating the Safety, Tolerability, Preliminary Efficacy, Pharmacokinetics, and Impact on Biomarkers of IPG11406 in Patients With Lupus Nephritis
Brief Title: Phase IIa Study for IPG11406 in Patients With Lupus Nephritis
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nanjing Immunophage Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IPG11406-C002
Record Dates: First submitted 2024-11-26; First posted 2024-12-05 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Lupus Nephritis
MeSH Terms: conditions — Lupus Nephritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (20 mg, Bid) (Experimental): 9~12 subjects will be orally administered with IPD11406 20 mg twice a day. All subjects will undergo screening for 28 days before administration, and those who pass the screening will undergo 28 days of drug administration and observation.
  Interventions: Drug: IPG11406
- Cohort 2 (40 mg, Bid) (Experimental): After cohort 1 complete 28 days of dosing and evaluation, the Safety Monitoring Committee (SMC) will assess the safety and tolerability of IPG11406 based on all accumulated safety data (including follow-up data) and available pharmacokinetic (PK) data. Based on SMC approval, 9~12 subjects will be orally administered 40 mg with IPD11406 twice a day. All subjects will undergo screening for 28 days before administration, and those who pass the screening will undergo 28 days of drug administration and observation.
  Interventions: Drug: IPG11406
- Cohort 3 (80 mg, Bid) (Experimental): After cohort 2 complete 28 days of dosing and evaluation, the Safety Monitoring Committee (SMC) will assess the safety and tolerability of IPG11406 based on all accumulated safety data (including follow-up data) and available pharmacokinetic (PK) data. Based on SMC approval, 9~12 subjects will be orally administered 80 mg with IPD11406 twice a day. All subjects will undergo screening for 28 days before administration, and those who pass the screening will undergo 28 days of drug administration and observation.
  Interventions: Drug: IPG11406

INTERVENTIONS:
Drug: IPG11406 — Investigational Medical Products:
  IPG11406 Activity: An antagonist of the GPR183 Dosage form: Tablet Strength: 10 mg and 40 mg Storage：15 ~ 25 °C in a tightly sealed container, protect from light Administration: In each cohort, IPG11406 tablets are orally administered twice a Day with an interval of 12±1 hours. Tablets should not be chewed or crushed.

SUMMARY:
A multi-center, multi-dose phase Ib/IIa clinical study evaluating the safety, tolerability, preliminary efficacy, pharmacokinetics, and impact on biomarkers of IPG11406 in patients with Lupus Nephritis

DETAILED DESCRIPTION:
This is a multi-center, multi-dose phase Ib/IIa study to evaluate the safety, tolerability, preliminary efficacy, pharmacokinetics, and impact on biomarkers of IPG11406 in patients with Lupus Nephritis.

Part A Three dose groups will be administered with drugs, namely 20 mg bid (cohort 1), 40 mg bid (cohort 2), and 80 mg bid (cohort 3). In cohorts 1 to 3, there will be 9-12 subjects in each cohort. All subjects will undergo screening for 28 days before administration, and those who pass the screening will undergo 28 days of drug administration and observation. This part plans to recruit about 36 patients with Lupus Nephritis.

After each cohort completes 28 days of dosing and evaluation, the Safety Monitoring Committee (SMC) will assess the safety and tolerability of IPG11406 based on all accumulated safety data (including follow-up data) and available pharmacokinetic (PK) data under blinded conditions. Based on the results of the safety and tolerability assessment, the SMC will decide whether to proceed with dosing in the next dose cohort. Part A will determine the recommended phase II dose (RP2D) and maximum tolerated dose (MTD) of IPG11406.

Part B The design of Part B will be finalized based on the results of Part A.

ELIGIBILITY:
Criteria for Inclusion and Exclusion <Inclusion Criteria>

1. The age range is between 18 and 70 years old (including 18 and 70), with no gender restrictions.
2. Weight ≥ 45kg.
3. Adult subjects who meet the revised classification criteria of the American College of Rheumatology (ACR) 1997 and were diagnosed with systemic lupus erythematosus before screening.
4. During the screening period, the disease activity was confirmed as follows: SLEDAI-2K score ≥ 6 points. Accompanied by lupus nephritis (according to the 2003 International Society of Nephrology/Renal Pathology Society (ISN/RPS) classification criteria, there is active, biopsy-confirmed type III or type IV proliferative lupus nephritis, with coexistence of type V allowed; the biopsy must be performed within 1 year before the screening visit or during the screening period, and the biopsy report is used to confirm patient eligibility.)
5. During the screening period, the patient's 24-hour urinary protein to creatinine ratio (UPCR) is greater than 1.0g/g, and the estimated glomerular filtration rate (eGFR) calculated using the MDRD formula is ≥60 mL/min/1.73 m^2; and the 24-hour urinary protein is ≥1g.
6. The patient's baseline serum IFN-γ exceeded the upper limit of normal values.
7. The Th1/Th2 ratio in peripheral blood of the patient during the baseline period is ≥14.
8. Subjects who have not undergone induction therapy are allowed to be enrolled, but during the study and follow-up period, they must not receive any other treatment for systemic lupus erythematosus and lupus nephritis. Subjects are allowed to be enrolled while receiving any of the following standard treatment regimens: 1) Oral prednisone (or equivalent) monotherapy: a. Treatment duration: medication use ≥2 weeks before screening and maintaining a stable dose ≥2 weeks before enrollment; b. Dose requirements: maximum daily dose: 1mg/kg/day; 2) Immunosuppressants: a. Permissible drugs include: antimalarials, azathioprine, cyclophosphamide, mycophenolate mofetil/mycophenolic acid, methotrexate, cyclosporine A, tacrolimus; b. Treatment duration: medication use ≥12 weeks before screening and maintaining a stable dose ≥8 weeks before enrollment; c. Dose requirements: hydroxychloroquine ≤400mg/day, azathioprine ≤100mg/day, cyclophosphamide ≤800mg/4 weeks, mycophenolate mofetil/mycophenolic acid ≤2g/day, oral, subcutaneous (SC), or intramuscular methotrexate ≤15mg/week, Cyclosporine A ≤ 3 mg/kg/d, tacrolimus ≤ 3 mg/d; 3) Oral prednisone (or equivalent medication) monotherapy ± hydroxychloroquine sulfate ± an immunosuppressant: a. The treatment duration and dose stability requirements for Oral glucocorticoids (OCS) and immunosuppressants mentioned above must be met; b. The maximum daily/weekly dose of each drug in 1) and 2) must not be exceeded.
9. Female subjects must be in a non-pregnant and non-breastfeeding period during the trial.
10. The subjects have no plans to become pregnant within 6 months after the screening and the end of the trial, voluntarily adopt effective contraceptive measures, and have no plans to donate sperm or eggs;
11. The subjects voluntarily participate in the study, are able to sign the informed consent form, and comply with the requirements stated on the informed consent form.

<Exclusion Criteria>

1. Pregnant and lactating women.
2. Screening for participation in other clinical trials within the previous 3 months and/or currently (excluding those who have not used the trial medication).
3. Active severe lupus nephritis, with estimated glomerular filtration rate (eGFR) calculated using the MDRD formula <60ml/min/1.73m^2.
4. Severe neuropsychiatric SLE includes but is not limited to the following: seizures, new or worsening impaired level of consciousness, psychosis, delirium or confusion state, aseptic meningitis, ascending or transverse myelitis, chorea, cerebellar ataxia, multiple mononeuropathy, demyelinating syndrome, or situations that make the subject unable to fully understand the ICF.
5. History or current diagnosis of clinically significant non-SLE-related vasculitis syndrome or overlap with other connective tissue diseases.
6. Any active skin diseases that may interfere with the research evaluation of SLE, including but not limited to psoriasis, dermatomyositis, systemic sclerosis, non-SLE skin lupus manifestations (such as skin vascular disease, perifollicular telangiectasia, fingertip sclerosis, rheumatoid nodules, erythema multiforme, leg ulcers) or drug-induced lupus, except for SLE.
7. Those with a history of lymphoproliferative diseases, or those who have had or currently have malignant tumors within the past 5 years (except for squamous cell carcinoma in situ, basal cell carcinoma, and cervical carcinoma in situ, which have been thoroughly treated and show no evidence of recurrence).
8. Patients with uncontrolled antiphospholipid syndrome (APS).
9. History of significant organ transplantation (e.g., heart, lung, kidney, liver) or hematopoietic stem cell/bone marrow transplantation.
10. Major surgical procedures (craniotomy, thoracotomy, or abdominal surgery) or unhealed wounds, ulcers, or fractures within 4 weeks before screening.
11. Individuals who have received live/attenuated vaccine within the 8 weeks before screening or plan to receive live/attenuated vaccine during the trial period.
12. Allergic to the trial medication (including excipients) or suffering from severe allergic diseases or belonging to an allergic constitution (such as being allergic to two or more drugs, foods, or pollen), which, in the judgment of the researcher, may compromise the safety of the subject.
13. During screening, any of the following cardiac impairments is present: a. New York Heart Association (NYHA) functional class III to IV; b. Uncontrolled angina, congestive heart failure, or myocardial infarction within 6 months prior to the first dose of medication; c. Prolonged QTcF interval calculated using the Fridericia formula (male > 450 msec; female > 470 msec); d. Second-degree type II atrioventricular (AV) block, third-degree AV block, or PR interval >250 msec; e. Various factors that may increase the risk of QTcF prolongation or arrhythmic events, such as heart failure, hypokalemia, congenital long QT syndrome, or a family history of sudden unexplained death of a first-degree relative before the age of 40; f. Left ventricular ejection fraction (LVEF) < 50%;
14. Active or latent tuberculosis infection during screening.
15. There is a serious herpes virus infection during screening, such as herpes encephalitis, disseminated herpes, and ocular herpes.
16. Needs to take oral anti-infective drugs (including antiviral drugs) or intravenous antibiotics due to infection within 2 weeks before screening.
17. Hospitalization due to opportunistic infections within 3 months before screening.
18. Treatment with traditional Chinese patent medicines and simple preparations such as Tripterygium Wilfordii within 4 weeks before screening.
19. Hepatitis B test shows HBsAg positive (if HBsAg is negative but HBcAb is positive, then HBV-DNA quantitative test is required, and patients with HBV-DNA test results ≥ the upper limit of the reference value of each center or requiring antiviral treatment do not meet the conditions to participate in the study), hepatitis C antibody positive (HCV-RNA test can be added, if negative, the patient can be included), Treponema pallidum antibody positive (if Treponema pallidum antibody is positive, further Treponema pallidum serological tests will be conducted. Patients who have been judged by the investigator to have been infected with syphilis in the past but have been cured meet the inclusion criteria), HIV antibody test positive.
20. During screening, subjects with significant abnormalities in liver and kidney function tests and blood routine examination, including: alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) exceeding twice the upper limit of normal values, total serum bilirubin exceeding 1.5 times the upper limit of normal values; serum creatinine greater than 1.5 times the upper limit of normal values; hemoglobin <90g/L; white blood cell count <3.0×10^9/L, platelet count (PLT) <75×10^9/L; neutrophil count <1.0×10^9/L; other laboratory test results that may affect the subject's ability to complete the trial or interfere with the trial results as judged by the investigator.
21. Those who have difficulty swallowing.
22. History of drug addiction or drug abuse;
23. Those who have acute diseases before using the clinical trial drugs;
24. Other conditions that the investigator deem unsuitable for enrollment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2026-04-22 (Estimated); Study Completion 2026-04-22 (Estimated)

PRIMARY OUTCOMES:
Evaluate the safety and tolerability via assessment of Adverse events | Up to 58 days
  Grades of AE will be assessed according to CTCAE 5.0
Evaluate the safety and tolerability via Respiration rate of Vital Signs | Up to 58 days
  Changes from baseline， Respiration rate in times per minute
Evaluate the safety and tolerability via Heart rate of Vital Signs | Up to 58 days
  Changes from baseline， Heart rate in beats per minute
Evaluate the safety and tolerability via Blood pressure of Vital Signs | Up to 58 days
  Changes from baseline，Blood pressure in mmHg
Evaluate the safety and tolerability via Body temperature of Vital Signs | Up to 58 days
  Changes from baseline，Body temperature in Celsius degree
Evaluating the safety and tolerability from Red blood cell count of Laboratory Examination | Up to 58 days
  Changes from baseline of Red blood cell count in whole blood is reported in the form of number.
Evaluating the safety and tolerability from White blood cell of Laboratory Examination | Up to 58 days
  Changes from baseline of White blood cell count in whole blood is reported in the form of number.
Evaluating the safety and tolerability from lymphocyte count of Laboratory Examination | Up to 58 days
  Changes from baseline , Lymphocyte count in whole blood is reported in the form of number.
Evaluating the safety and tolerability from hemoglobin of Laboratory Examination | Up to 58 days
  Changes from baseline , Changes of hemoglobin concentration（g/dL）in whole blood will be recorded.
Evaluating the safety and tolerability from Laboratory Examination | Up to 58 days
  Changes from baseline of Laboratory Examination (hematology, clinical chemistry, coagulation, urinalysis)
Evaluating the safety and tolerability from Prothrombin time of Laboratory Examination | Up to 58 days
  Changes from baseline, Prothrombin time (PT) is a screening test for exogenous coagulation factors.
Evaluating the safety and tolerability from Activated partial thromboplastin time of Laboratory Examination | Up to 58 days
  Changes from baseline, Activated partial thromboplastin time (APTT) is a screening test for endogenous coagulation factors.
Evaluating the safety and tolerability from total bilirubin concentration of Laboratory Examination | Up to 58 days
  Changes from baseline, Changes of total bilirubin concentration (μmol/L) in serum will be recorded.
Evaluating the safety and tolerability from direct bilirubin concentratio of Laboratory Examination | Up to 58 days
  Changes from baseline, Changes of direct bilirubin concentration (μmol/L) in serum will be recorded.
Evaluating the safety and tolerability from ALT of Laboratory Examination | Up to 58 days
  Changes from baseline, Changes of ALT concentration (U/L) in serum will be recorded.
Evaluating the safety and tolerability from AST of Laboratory Examination | Up to 58 days
  Changes from baseline, Changes of AST concentration (U/L) in serum will be recorded.
Evaluating the safety and tolerability from creatinine concentration of Laboratory Examination | Up to 58 days
  Changes from baseline, Changes of creatinine concentration (μmol/L) in serum will be recorded.
Evaluating the safety and tolerability from triglyceridesconcentration of Laboratory Examination | Up to 58 days
  Changes from baseline, Changes of triglycerides (TG) concentration (mmol/L) in serum will be recorded.
Evaluating the safety and tolerability from urine protein of Laboratory Examination | Up to 58 days
  Changes from baseline, Changes of urine protein will be examined by qualitative test
Evaluating the safety and tolerability from urine pH value of Laboratory Examination | Up to 58 days
  Changes from baseline, Changes of urine pH value will be recorded.
Evaluating the safety and tolerability from ventricular rate of Electrocardiogram | Up to 58 days
  Changes from Clinical Significant Changes in 12-Lead Electrocardiogram (ECG) findings for ventricular rate (beats/min)
Evaluating the safety and tolerability from PR interval of Electrocardiogram | Up to 58 days
  Changes from Clinical Significant Changes in 12-Lead Electrocardiogram (ECG) findings for PR interval (ms)
Evaluating the safety and tolerability from QRS (ms) of Electrocardiogram | Up to 58 days
  Changes from Clinical Significant Changes in 12-Lead Electrocardiogram (ECG) findings for QRS (ms)
Evaluating the safety and tolerability from QTc of Electrocardiogram | Up to 58 days
  Changes from Clinical Significant Changes in 12-Lead Electrocardiogram (ECG) findings for QTc (ms),
Evaluate the impact of oral IPG11406 on biomarkers in patients with Lupus Nephritis | Up to 58 days
  Changes in biomarkers before and after medication administration in patients
Evaluate the impact of oral administration of IPG11406 on 24-hour urine protein quantitation of proteinuria and renal function in patients with Lupus Nephritis | Up to 58 days
  Measure the changes in 24-hour urine protein quantitation before and after medication administration
Evaluate the impact of oral administration of IPG11406 on estimated glomerular filtration rate of proteinuria and renal function in patients with Lupus Nephritis | Up to 58 days
  Measure the changes in estimated glomerular filtration rate (eGFR) calculated using the MDRD formula before and after medication administration
Evaluate the impact of oral administration of IPG11406 on ratio of 24-hour urine protein to urine creatinine of proteinuria and renal function in patients with Lupus Nephritis | Up to 58 days
  Measure the changes in ratio of 24-hour urine protein to urine creatinine before and after medication administration
Evaluate the impact of oral administration of IPG11406 on proteinuria and renal function in patients with Lupus Nephritis | Up to 58 days
  Measure the changes in 24-hour urine protein quantitation, estimated glomerular filtration rate (eGFR) calculated using the MDRD formula, and the ratio of 24-hour urine protein to urine creatinine before and after medication administration

SECONDARY OUTCOMES:
Evaluate the pharmacokinetics (PK) characteristics of oral IPG11406 in Maximum Plasma Concentration | Up to 28 days
  PK parameters:Maximum Plasma Concentration [Cmax]
Evaluate the pharmacokinetics (PK) characteristics of oral IPG11406 in Area under the curve | Up to 28 days
  PK parameters (under food effect): Area Under The Curve (AUC)
Evaluate the pharmacokinetics (PK) characteristics of oral IPG11406 from clearance at steady state | Up to 28 days
  PK parameters (under food effect): clearance at steady state (CLss/F)
Evaluate the pharmacokinetics (PK) characteristics of oral IPG11406 from T1/2 | Up to 28 days
  Elimination half-life (T1/2) after dose
Evaluate the pharmacokinetics (PK) characteristics of oral IPG11406 in CL by plasma concentration of whole blood sample | Up to 28 days
  Clearance (CL) after dose
Evaluate the preliminary efficacy of oral IPG11406 from peripheral blood T lymphocyte counts and proportion | Up to 58 days
  Changes in peripheral blood T lymphocyte counts and proportions before and after medication administration
Evaluate the preliminary efficacy of oral IPG11406 from Autoantibodies | Up to 58 days
  Changes in autoantibodies before and after medication administration
Evaluate the preliminary efficacy of oral IPG11406 from Relative count of lymphocyte subsets | Up to 58 days
  Changes in Relative count of lymphocyte subsets before and after medication administration
Evaluate the preliminary efficacy of oral IPG11406 from cytokines | Up to 58 days
  Changes in cytokines before and after medication administration
Evaluate the preliminary efficacy of oral IPG11406 from Th1/Th2 detection | Up to 58 days
  Changes in Th1/Th2 before and after medication administration
Evaluate the preliminary efficacy of oral IPG11406 from Routine immunological tests | Up to 58 days
  Changes in Routine immunological tests before and after medication administration
Evaluate the preliminary efficacy of oral IPG11406 in patients with Lupus Nephritis | Up to 58 days
  Changes in peripheral blood B lymphocyte and T lymphocyte counts and proportions, serum albumin, blood creatinine, blood uric acid, blood urea nitrogen (BUN), white blood cells, blood neutrophils, C-reactive protein, complement C3, complement C4, immunoglobulins (IgG, IgA, IgM, IgE), anti-ds-DNA antibody, anti-nuclear antibody, anti-cardiolipin antibody (A/G/M, IgG, IgM), anti-histone antibody, anti-nucleosome antibody, anti-ribosomal P protein antibody, anti-sm antibody, anti-SSA antibody, IL-6, IL-17, IL-2, IL-1β, IL-10, IFN-α, TNF-α, ferritin, and SLEDAI-2K score before and after medication administration
Evaluate the preliminary efficacy of oral IPG11406 from tests from antiphospholipid antibodies | Up to 58 days
  Changes in tests for antiphospholipid antibodies before and after medication administration
Evaluate the preliminary efficacy of oral IPG11406 from 24-hour urine protein test | Up to 58 days
  Changes in 24-hour urine protein test before and after medication administration
Evaluate the preliminary efficacy of oral IPG11406 from Serum ferritin | Up to 58 days
  Changes in Serum ferritin before and after medication administration
Evaluate the preliminary efficacy of oral IPG11406 from Systemic Lupus Erythematosus Disease Activity Index 2000（SLEDAI-2K） score | Up to 58 days
  Changes in SLEDAI-2K score before and after medication administration。
  Minimum and Maximum Values:
  The SLEDAI-2K score ranges from 0 (indicating no disease activity) to a maximum possible score that depends on the specific items being scored. However, in practical clinical use, the maximum score is typically much lower than the theoretical maximum, as not all items will be positive in any given patient. The exact maximum score can vary slightly depending on the specific version of the SLEDAI-2K being used, but it is generally well below 100.
  In the SLEDAI-2K, higher scores indicate a worse outcome. This is because the scale assigns points based on the presence and severity of various lupus manifestations, such as arthritis, rash, fever, and organ involvement. Therefore, as the score increases, it reflects greater disease activity and potentially more severe disease manifestations.

CONTACTS AND LOCATIONS:
Locations (17):
- China (17):
  - The First Affiliated Hospital Of Anhui Medical University, Hefei, Anhui
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Fujian Provincial Hospital, Fuzhou, Fujian
  - Sun Yai-sen Memorial Hospital, Sun Yai-sen University, Guangzhou, Guandong
  - Hebei Petro China Central Hospital, Langfang, Hebei
  - Xinxiang Central Hospital, Xinxiang, Henan
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Wuhan Hospital of Traditional Chinese and Western Medicine, Wuhan, Hubei
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - Nanjing DrumTower Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - Nantong First People's Hospital, Nantong, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Shandong Provincial Hospital, Jinan, Shandong
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Jinhua Municipal Centeral Hospital Medical Group, Jinhua, Zhejiang

IPD SHARING:
Plan to Share IPD: No